CLINICAL TRIAL: NCT04368871
Title: Radiographic Findings and Their Temporal Changes in COVID-19 Positive Changes Patients: A Prospective Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Max Healthcare Insititute Limited (Other)
Responsible Party: Sponsor
Other Study IDs: Covid-19/RFTC/MHC/2020
Record Dates: First submitted 2020-04-29; First posted 2020-04-30 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-04

CONDITIONS: COVID

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
All Patient irrespective of age with confirmed COVID-19 admitted to hospital and who underwent chest radiograph will be enrolled in the study to find raduigraphic findings and their temporal changes in COVID-19.

DETAILED DESCRIPTION:
In this prospective trial the investigator will work on radiology findings and their temporal changes in COVID-19 positive patients and who underwent chest radiograph will be enrolled in our study.

Patient selection will be consecutive in addition of age , gender and comorbid conditions clinical information will included travel,expose and contact history. All patients should be positive for COVID-19 via laboratory testing with real time reverse transcriptase polymerase chain reaction(rRT-PCR) In addition, the number of rRT-PCR tests performed on each patient, on which test a positive result was found,and the number of days between symptomology onset and date of first positive test will be recorded.

In view of the current dynamics, any other reliable diagnostic test(s) if added to the clinical protocol will also be considered for inclusion in this study.

Tabulation of radiographic findings for all consecutive X-rays will be done along with the temporal changes of these findings. further, the clinical findings with the outcomes(duration of hospital findings, ventilatory support and discharge/death).

ELIGIBILITY:
Inclusion Criteria:

1.Patients confirmed positive for COVID-19 by rRT-PCR irrespective of age.

Exclusion Criteria:

1.Patients with flu like symptoms but negative for COVID-19 by rRT-PCR.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: the study population will include all the COVID-19 pateints of Max Super speciality Hospital, New Delhi, India, all males and females with minimum age 18 years old and who underwent Chest radiograph will be included in the study
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-04-28 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
Radiographic findings and their temporal changes in COVID-19 positive patient: A Prospective study | 1-2 weeks
  Determine the radiographic findings in chest X-ray of COVID-19 positive patients.

SECONDARY OUTCOMES:
Radiographic findings and their temporal changes in COVID-19 positive patient: A Prospective study | 4-8 weeks
  Correlation of clinical findings with the outcomes (duration of hospital stay, ventilatory support, and discharge/death)

CONTACTS AND LOCATIONS:
Locations (1):
- Max Super Speciality Hospital, A Unit of Devki Devi Foundation, New Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided
IPD sharing protocol is undecided at this stage. We may, however, provide data if required